CLINICAL TRIAL: NCT04064619
Title: Recurrence of Symptoms of Overactive Bladder After Weaning Versus Sudden Stopping of Anticholinergics
Brief Title: Compare Sudden Stopping and Weaning of Anticholinergics in Recurrence of OAB Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed M Abdelbary, MD, Associate professor, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anticholinergic weaning
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Voiding Disorders
Keywords: OAB
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Intervention Model Description: 60 patients with idiopathic OAB and treated with solifenacin 5mg twice daily for one month. After improvement of their condition, we divided the responders into 2 groups, group I stopped the drug suddenly, while group II underwent gradual weaning of the drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sudden stopping (Active Comparator): patients were followed up after 1 and 3 months from stopping the drug,
  Interventions: Drug: Solifenacin Succinate 5 MG
- Weaning (Experimental): patients were followed up after 1and 3 months from the end of gradual weaning
  Interventions: Drug: Solifenacin Succinate 5 MG

INTERVENTIONS:
Drug: Solifenacin Succinate 5 MG — gradual weaning of drug vs. stopping
  Other Names: vesicare

SUMMARY:
Our study included 60 patients with idiopathic OAB and treated with solifenacin 5mg twice daily for one month. After improvement of their condition, we divided the responders into 2 groups, group I stopped the drug suddenly, while group II underwent gradual weaning of the drug.

DETAILED DESCRIPTION:
We started an open-label, prospective, two-arm, randomized controlled trial at Beni-Suef University, from January 2018 to January 2019, including 60 patients suffering from OAB symptoms. Patients were recently diagnosed with idiopathic OAB which was not treated prior to enrollment. All participants signed written informed consents. The study protocol was approved by the ethics committee of our faculty. Patients were allocated into 2 equal groups (30 patients in each group) according to a computer-generated random numeric table after exclusion of those who are not eligible or refused to be included in the study

ELIGIBILITY:
Inclusion Criteria:

* OAB patients.
* Recently diagnosed.

Exclusion Criteria:

* Previous trials of treatment
* UTI, stones, tumors, or Infravesical obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
improvement | 1 month
  decrease voiding times

SECONDARY OUTCOMES:
recurrence of symptoms | 3 months
  increase in voiding times after improvement

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelbary, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No